CLINICAL TRIAL: NCT01628536
Title: A Pilot Pre-operative Window Trial of Black Cohosh in Women With Ductal Carcinoma in Situ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1205010204
Record Dates: First submitted 2012-06-20; First posted 2012-06-26 (Estimated); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Ductal Carcinoma in Situ
Keywords: Black Cohosh; Ductal Carcinoma in situ; Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms | interventions — black cohosh root extract; Remifemin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Black cohosh (Experimental)
  Interventions: Dietary Supplement: Black cohosh

INTERVENTIONS:
Dietary Supplement: Black cohosh — Remifemin 20 mg tablet orally twice per day x 4 weeks
  Other Names: Remifemin

SUMMARY:
The investigators hypothesize that black cohosh, as a potentially therapeutic agent, will reduce the overall size and aggressiveness of ductal carcinoma in situ (DCIS) when given in a pre-operative setting.

DETAILED DESCRIPTION:
The overarching hypothesis of our research is that black cohosh has potential to be a well-tolerated, effective agent for the treatment of early breast cancer. This pilot study represents a first step in exploring this hypothesis by demonstrating preliminary evidence of specific anti-tumor effect of black cohosh on areas of ductal carcinoma in situ (DCIS) in the breast.

ELIGIBILITY:
Inclusion Criteria:

* A patient/subject is eligible for enrollment if all of the following inclusion criteria are met:

  1. Pre- and post-menopausal women ≥ 18 years of age newly diagnosed with DCIS histologically confirmed on breast core biopsy
  2. Ability to understand and the willingness to sign a written informed consent document
  3. ECOG performance status 0-1
  4. Life expectancy >12 months
  5. Willing to schedule definitive resection of DCIS 4 weeks +/- 1 week after study enrollment
  6. Original breast core biopsy specimen available for pathologic review and staining by Yale School of Medicine Department of Pathology

Exclusion Criteria:

* A patient /subject will not be eligible for this study if any of the following exclusion criteria are met:

  1. Pregnant or nursing within past 6 months
  2. Lactose intolerant, lactose allergy or salicylate allergy
  3. Patients who have already undergone excisional biopsy for qualifying DCIS
  4. Patients with ipsilateral treatment for DCIS or breast cancer within 12 months prior to entering this study
  5. Patients receiving any other chemotherapy or investigational agents
  6. Serious concomitant systemic disorders (including active infections) or psychiatric illness/social situations that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
  7. Liver function tests ≥ 20% of the institutional upper limits of normal
  8. Creatinine > 1.5 times the institutional upper limit of normal
  9. ANC < 1,500 /µL
  10. Platelets < 100,000 /µL
  11. History of allergic reactions attributed to compounds of similar chemical or biologic composition to black cohosh
  12. The effects of black cohosh on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
  13. Prior/concurrent therapy including:

      Tamoxifen, raloxifene, letrozole, anastrozole, or exemestane in the past 6 months
  14. Chemotherapy, biologic therapy (e.g., trastuzumab [Herceptin®]), or breast radiotherapy to the breast currently affected by DCIS within the past 12 months
  15. Any exogenous hormonal therapy including estrogen-, progesterone-, and/or androgen-based agents in the past 6 months
  16. Phytoestrogens or OTC medications with estrogenic or androgenic properties in the past 6 months
  17. Any black cohosh preparation within the past 6 months

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-06; Primary Completion 2016-01-14 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Measure change in size of DCIS on routine imaging | 4 weeks
  1. Measure change in size of DCIS on routine imaging (i.e. mammography and/or ultrasound) obtained before and after 4 weeks of treatment with black cohosh, with correlation to specimen sizes; and
  2. Determine differences in breast epithelial cell proliferation in areas of DCIS as measured by mean change in levels of Ki67 before and after 4 weeks of treatment with black cohosh. Ki67 levels will be assessed with traditional immunohistochemical staining as well as AQUA technology.

SECONDARY OUTCOMES:
Assess adherence to a brief course of black cohosh. | 4 weeks
  To test this secondary hypothesis, we will:
  Assess adherence to a brief course of black cohosh. Participants will be given an adequate supply of medication for 4 weeks +/- 1 week at the screening/enrollment visit. They will be instructed to bring their medication back on the day of surgery. Pill counts will be conducted by the research nurse to assess the participant's level of compliance.
Assess safety and side effects of 4 week course of black cohosh | 4 weeks
  To assess this secondary outcome measure we will:
  Assess safety and side effects through patient history, pill diary and safety labs.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Hofstatter, MD, Principal Investigator — Yale University
Locations (1):
- Erin Hofstatter, MD, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Trant AA, Chagpar A, Wei W, Neumeister V, Rimm D, Stavris K, Lurie B, Frederick C, Andrejeva L, Raghu M, Killelea B, Horowitz N, Lannin D, Knill-Selby E, Sturrock T, Hofstatter E. The Effect of Black Cohosh on Ki67 expression and Tumor Volume: A Pilot Study of Ductal Carcinoma in Situ Patients. Integr Cancer Ther. 2022 Jan-Dec;21:15347354221137290. doi: 10.1177/15347354221137290. PMID 36444764
- See also: Yale Cancer Center Studies — http://www.yalestudies.org